CLINICAL TRIAL: NCT02441049
Title: Latino Mothers as Primary Agents of Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: San Diego State University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Guadalupe X. Ayala, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G00007105
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Eating Behavior
Keywords: Latino; Hispanic; Diet; Family health; Promotora; Intervention
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home-based promotora intervention (Experimental): Study participants and their families received the home-based promotora family intervention
  Interventions: Behavioral: Home-based promotora family intervention
- Delayed treatment control (No Intervention): Study participants received intervention materials after the final study evaluation measures were taken, 10 months post-baseline.

INTERVENTIONS:
Behavioral: Home-based promotora family intervention — A promotora-delivered family intervention in the participant's home. Promotoras used a telenovela-style DVD and accompanying manual to deliver 11 home sessions to the family, and 4 support telephone calls, over a 4 month period.
  Other Names: Entre Familia: Reflejos de Salud
  Arms: Home-based promotora intervention

SUMMARY:
Entre Familia was a 4-year randomized controlled trial funded by the American Cancer Society. The study was conducted in Imperial County, California, and involved a partnership between the Institute for Behavioral and Community Health at San Diego State University and Clínicas de Salud del Pueblo, Inc. a private, non-profit corporation providing comprehensive primary care services to residents throughout Imperial and Riverside Counties. The investigators enrolled 361 Latina mothers and one of their children aged between 7 and 13 years old; in 25% of families, the father was also enrolled. Participants were randomly assigned to either an intervention or delayed-treatment control condition. The intervention consisted of a community health worker (or promotora)-delivered home-based intervention to promote healthy eating. The promotoras used a telenovela DVD series and accompanying manual, both written and produced by study staff. The intervention was delivered through 11 home visits and 4 support telephone calls over a 4 month period. Participants in the delayed-treatment condition received intervention materials when evaluation assessments had been completed. Evaluation measures were taken at baseline, 4 months (immediate post-intervention) and 10 months (6-months post intervention). Participants completed a self-report interview with study staff at each time point. Height and weight measurements were also collected for the mothers and children. The primary outcomes were changes in mothers' daily fruit and vegetable intake. Secondary outcomes for mothers, children and fathers included changes in fat intake, sugary beverage intake, parenting strategies, and perceived barriers to healthy eating.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* must self-identify as Latina,
* must be able to read and speak Spanish,
* must be at least 18 years old,
* must be a resident of Imperial County,
* and must plan to reside in the county for the 10 month study duration.

Children (both genders):

* must be between the ages of 7-13 years,
* must reside with his/her mother and her spouse/partner for at least 4 days of the week.

Exclusion Criteria:

* Families who intend to move away from Imperial County before the end of the study, and families with a family member on a medically-prescribed diet

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in mother daily fruit and vegetable intake in the past month between baseline, immediate-post intervention and 6-months post-intervention, assessed using the NCI Fruit and Vegetable All-Day Screener | Baseline, 4 months, 10 months

SECONDARY OUTCOMES:
Child, father: change in daily fruit and vegetable intake in the past month between baseline, immediate-post intervention and 6-months post-intervention, assessed using the NCI Fruit and Vegetable All-Day Screener | Baseline, 4 months, 10 months
Mother, child, father: change in monthly fruit and vegetable variety between baseline, immediate-post intervention and 6-months post-intervention, assessed using self-reported intake of 32 fruits and 43 vegetables | Baseline, 4 months, 10 months
Mother, father: change in perceived quality of diet between baseline, immediate-post intervention and 6-months post-intervention, assessed using one item from the 2005-06 NHANES (Diet Behavior and Nutrition module) | Baseline, 4 months, 10 months
Mother, father: change in parenting strategies between baseline, immediate-post intervention and 6-months post-intervention, assessed using a modified version of the PEAS scale | Baseline, 4 months, 10 months
Mother: change in social support for fruit and vegetable intake between baseline, immediate-post intervention and 6-months post-intervention, assessed using a modified version of preexisting F&V shopping practices and social support scales | Baseline, 4 months, 10 months
Mother, child, father: change in weekly fast food intake between baseline, immediate-post intervention and 6-months post-intervention, assessed by asking for self-reported number of days in a typical week the respondent ate at fast food restaurants | Baseline, 4 months, 10 months
Mother, father: change in perceived barriers to obtaining and consuming fruits and vegetables between baseline, immediate-post intervention and 6-months post-intervention, assessed using 11-items including ease of purchasing F&V in the neighborhood | Baseline, 4 months, 10 months
Mother, father: change in fat intake between baseline, immediate-post intervention and 6-months post-intervention, assessed using the NCI Multifactor Fat Screener | Baseline, 4 months, 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe X Ayala, PhD, MPH, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University Research Foundation, San Diego, California, United States

REFERENCES:
- [Result] Horton LA, Parada H, Slymen DJ, Arredondo E, Ibarra L, Ayala GX. Targeting children's dietary behaviors in a family intervention: 'Entre familia: reflejos de salud'. Salud Publica Mex. 2013;55 Suppl 3:397-405. PMID 24643488
- [Result] Ayala GX, Ibarra L, Horton L, Arredondo EM, Slymen DJ, Engelberg M, Rock CL, Hernandez E, Parada H, Elder JP. Evidence supporting a promotora-delivered entertainment education intervention for improving mothers' dietary intake: the Entre Familia: Reflejos de Salud Study. J Health Commun. 2015;20(2):165-76. doi: 10.1080/10810730.2014.917747. Epub 2014 Nov 6. PMID 25375276
- [Result] Schmied E, Parada H, Horton L, Ibarra L, Ayala G. A Process Evaluation of an Efficacious Family-Based Intervention to Promote Healthy Eating: The Entre Familia: Reflejos de Salud Study. Health Educ Behav. 2015 Oct;42(5):583-92. doi: 10.1177/1090198115577375. Epub 2015 Mar 25. PMID 25810469
- [Result] Ayala, G.X., Ibarra, L., Arredondo, E., Horton, L., Hernandez, E., Parada, H., Slymen, D., Rock, C., Engelberg, M., Elder, J.P. (2011). Promoting healthy eating by strengthening family relations: Design and implementation of the Entre Familia: Reflejos de Salud intervention. In R. Elk & H. Landrine (Eds.), Cancer Disparities: Causes and Evidence-Based Solutions. Springer.
- [Result] Schmied EA, Parada H, Horton LA, Madanat H, Ayala GX. Family support is associated with behavioral strategies for healthy eating among Latinas. Health Educ Behav. 2014 Feb;41(1):34-41. doi: 10.1177/1090198113485754. Epub 2013 May 27. PMID 23711676
- [Result] Parada H, Ayala GX, Horton LA, Ibarra L, Arredondo EM. Latino fathers' feeding-related parenting strategies on children's eating. Ecol Food Nutr. 2016 May-Jun;55(3):292-307. doi: 10.1080/03670244.2016.1161616. Epub 2016 Apr 11. PMID 27065160
- [Result] Soto SC, Arredondo EM, Horton LA, Ayala GX. Validation of the modified Parenting Strategies for Eating and Physical Activity Scale-Diet (PEAS-Diet) in Latino children. Appetite. 2016 Mar 1;98:55-62. doi: 10.1016/j.appet.2015.12.003. Epub 2015 Dec 15. PMID 26699670
- [Derived] Arredondo EM, Ayala GX, Soto S, Slymen DJ, Horton LA, Parada H, Campbell N, Ibarra L, Engelberg M, Elder JP. Latina mothers as agents of change in children's eating habits: findings from the randomized controlled trial Entre Familia: Reflejos de Salud. Int J Behav Nutr Phys Act. 2018 Oct 1;15(1):95. doi: 10.1186/s12966-018-0714-0. PMID 30285755
- [Derived] Horton LA, Ayala GX, Slymen DJ, Ibarra L, Hernandez E, Parada H, Rock CL, Arredondo EM, Elder JP. A Mediation Analysis of Mothers' Dietary Intake: The Entre Familia: Reflejos de Salud Randomized Controlled Trial. Health Educ Behav. 2018 Aug;45(4):501-510. doi: 10.1177/1090198117742439. Epub 2017 Dec 6. PMID 29212358